CLINICAL TRIAL: NCT03115099
Title: A Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY3325656 After Single Dose in Healthy Subjects and Patients With Type 2 Diabetes
Brief Title: A Study of LY3325656 in Healthy Participants and Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16433; I8U-MC-DMBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo (Part A) (Placebo Comparator): Single oral dose of placebo (sugar pill) administered to healthy participants in up to 1 study period in Part A
  Interventions: Drug: Placebo
- LY3325656 (Part A) (Experimental): Single ascending dose of LY3325656 administered orally to healthy participants in up to 3 study periods in Part A
  Interventions: Drug: LY3325656
- Placebo (Part B) (Placebo Comparator): Single oral dose of placebo (sugar pill) administered to participants with T2DM in 1 study period in Part B
  Interventions: Drug: Placebo
- LY3325656 (Part B) (Experimental): Single oral dose of LY3325656 administered to participants with T2DM in 1 study period in Part B
  Interventions: Drug: LY3325656
- Liraglutide (Part B) (Active Comparator): Single subcutaneous dose of liraglutide administered to participants with T2DM in 1 study period in Part B
  Interventions: Drug: Liraglutide
- LY3325656 + Sitagliptin (Part B) (Experimental): Single oral dose of LY3325656 and sitagliptin administered to participants with T2DM in 1 study period in Part B
  Interventions: Drug: LY3325656; Drug: Sitagliptin

INTERVENTIONS:
Drug: LY3325656 — Administered orally
  Arms: LY3325656 (Part A); LY3325656 (Part B); LY3325656 + Sitagliptin (Part B)
Drug: Placebo — Administered orally
  Arms: Placebo (Part A); Placebo (Part B)
Drug: Liraglutide — Administered subcutaneously
  Arms: Liraglutide (Part B)
Drug: Sitagliptin — Administered orally
  Arms: LY3325656 + Sitagliptin (Part B)

SUMMARY:
The aim of this trial is to evaluate the safety of single doses of a study drug known as LY3325656 that is given orally to healthy participants and participants with type 2 diabetes. Information about any side effects that may occur will be collected.

It will also investigate how much of the study drug gets into the blood stream, and how long it takes the body to get rid of it.

The study consists of two parts. Part A will study healthy participants over approximately 12 weeks and Part B will study participants with type 2 diabetes over approximately 5 weeks, excluding screening. Screening is required within 28 days of the start of the study.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Must be a male, or a female who cannot become pregnant, and who is either a healthy participant, or who has type 2 diabetes
* Have a screening body mass index (BMI) of at least 18.5 kilograms per square meter (kg/m²)
* Have blood pressure, pulse rate, blood and urine laboratory test results acceptable for the study

For participants with Type 2 Diabetes Mellitus:

* Have diabetes controlled on diet and exercise with or without metformin for at least 30 days prior to screening, or on sulfonylureas with or without metformin
* Have a glycated hemoglobin (HbA1c) value of greater than or equal to 7% and less than or equal to 11% at screening (exercise with or without metformin)
* Have a HbA1c value of greater than or equal to 7% and less than or equal to 8.5% at screening (sulfonylureas with or without metformin)

Exclusion Criteria:

For all participants:

* Are currently participating in another clinical study or completed one in the last 30 days
* Are allergic to LY3325656 or other related drugs
* Have a history of significant heart, lung, liver, kidney, stomach or brain disease, or have any medical problems which may cause an increased risk during the study
* Have electrocardiogram (ECG) readings that are not suitable for the study
* Are infected with hepatitis B
* Are infected with human immunodeficiency virus (HIV)
* Have donated more than 450 mL of blood in the last 3 months or if have donated any blood in the last month
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female), or are unwilling to stop alcohol as required by the study restrictions (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of spirits)
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic

For participants with Type 2 Diabetes Mellitus:

* Have had heart disease or stroke within 6 months before entering the study
* Have health complications due to poorly controlled diabetes as shown by blood and urine laboratory test results or based on physical examination and medical assessment as determined by the study doctor
* Have been hospitalized for poor control of diabetes (keto-acidotic episode) in the last 6 months
* Have used insulin to control diabetes in the last 6 months
* Show symptoms of high blood sugar e.g. frequent urination, always feeling thirsty, or unexpected weight loss

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through approximately 12 weeks and 5 weeks after first administration of study drug in Parts A and B, respectively
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3325656 | Baseline up to 72 hours after each dose of study drug
  Pharmacokinetics: Area Under the Concentration Curve of LY3325656 From Time Zero to 24 Hours [AUC(0-24)]
Pharmacokinetics: Maximum Concentration (Cmax) of LY3325656 | Baseline up to 72 hours after each dose of study drug
  Pharmacokinetics: Maximum Concentration (Cmax) of LY3325656

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Singapore (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Singapore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore